CLINICAL TRIAL: NCT01365481
Title: A Multicenter, Open-label, 18 Month Study to Evaluate the Long-term Safety and Tolerability of Valsartan in Children 6 to 17 Years of Age With Hypertension and With or Without Chronic Kidney Disease
Brief Title: Safety and Tolerability of Valsartan in Children 6 to 17 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAL489K2305; 2009-017594-37 (EudraCT Number)
Record Dates: First submitted 2011-05-09; First posted 2011-06-03 (Estimated); Results first posted 2016-04-21 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-06

CONDITIONS: Hypertension; Chronic Kidney Disease
Keywords: Hypertension, pediatric; Hypertension with or without chronic kidney disease
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic | interventions — Valsartan; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- valsartan (Experimental): Valsartan starting dose: ≥18 kg to <35 kg is 40 mg, ≥35 kg to <80 kg is 80 mg, ≥80 kg to ≤160 kg is 160 mg for 1 week then Valsartan maintenance dose: ≥18 kg to <35 kg is 80 mg, ≥35 kg to <80 kg is 160 mg, ≥80 kg to ≤160 kg is 320 mg after Week 8 if the Mean Sitting Systolic Blood Pressure (MSSBP) and/or Mean Sitting Diastolic Blood Pressure (MSDBP) was higher than 95th percentile for age, gender and height under the maintenance valsartan dose then add amlodipine and/or Hydrochlorothiazide (HCTZ). The valsartan +antihypertensive group includes patients who received background antihypertensive medication or received antihypertensive medication including amlodipine or HCTZ during the study.
  Interventions: Drug: Valsartan; Drug: amlodipine; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Valsartan — week 1: 40/80/160 week 2-78: 80/160/320mg, oral, by mouth, once daily
  Other Names: VAL489
Drug: amlodipine — added to valsartan after week 8 if the MSSBP and/or MSDBP was higher than 95th percentile for age, gender and height under the maintenance valsartan dose
Drug: Hydrochlorothiazide — added to valsartan after week 8 if the MSSBP and/or MSDBP was higher than 95th percentile for age, gender and height under the maintenance valsartan dose
  Other Names: HCTZ

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability profile of valsartan and valsartan-based treatments in children with hypertension, with or without chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of hypertension
* able to swallow a tablet
* body weight ≥18 kg and ≤160 kg at baseline
* MSSBP must be ≥ 95th percentile and ≤25% above the 95th percentile for age, gender and height.

Exclusion Criteria:

* Any clinically significant physical abnormalities or clinically relevant abnormal laboratory values (other than those relating to renal function) obtained at the screening visit. Including the following:

  1. AST/SGOT or ALT/SGPT >3 times the upper limit of the reference range. Patients known to have active or chronic hepatitis were excluded.
  2. Total bilirubin >2 times the upper limit of the reference range
  3. Estimated GFR <30 mL/min/1.73m² (calculated using Modified Schwartz Formula)
  4. WBC count <3000/mm³
  5. Platelet count <100,000/mm³
  6. Serum potassium >5.3 mmol/L
  7. Hemoglobin <8 g/dL
* Uncontrolled diabetes mellitus
* Unilateral, bilateral and graft renal artery stenosis
* Current diagnosis of heart failure (New York Heart Association Class II-IV)
* Patients taking any of the following concomitant medications following screening: Renin-angiotensin receptor(RAAS) blockers other than study drug, Lithium, potassium-sparing diuretics, potassium supplements, salt substitutes containing potassium and other substances that may increase potassium levels, Non-steroidal anti-inflammatory drugs (NSAIDS), including selective COX-2 inhibitors, acetylsalicylic acid >3g/day, and non-selective NSAIDs, Antidepressant drugs in the class of Monoamine oxidase (MAO) inhibitors (e.g. phenelzine), Chronic use of stimulant therapy for Attention deficit disorder/attention deficit hyperactivity disorder (ADD/ADHD) -Patients who demonstrate clinically significant ECG abnormalities such as concurrent potentially life threatening arrhythmia or symptomatic arrhythmia and patients with second or third degree heart block without a pacemaker.
* Coarctation of the aorta with a gradient of >=30 mmHg
* Previous solid organ transplantation except renal transplantation.
* Patients known to be positive for the human immunodeficiency virus (HIV)
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of the study drug
* Known or suspected contraindications to the study drug, including severe hepatic impairment, biliary cirrhosis, cholestasis and history of allergy to ARBs and/or angiotensin-converting enzymes (ACE) and/or Direct Renin Inhibitors (DRIs)
* History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
* History or evidence of drug or alcohol abuse within the last 12 months.
* Female patients of child-bearing potential, defined as all female patients physiologically capable of becoming pregnant, unless they are willing to use highly effective contraception during the study
* Pregnant or nursing (lactating) female patients
* Participation in any investigational drug study within 30 days prior to screening or within 5 elimination half-lives of the study drug prior to screening, or whichever is longer.
* History of hypersensitivity to the study drug or to drugs of similar chemical classes.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2011-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- Colombia (3):
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Cali
- Novartis Investigative Site, Helsinki, Finland, Finland
- Germany (5):
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Cottbus
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Rostock
- Novartis Investigative Site, Guatemala City, Departamento de Guatemala, Guatemala
- Philippines (2):
  - Novartis Investigative Site, Manila, Philippines
  - Novartis Investigative Site, Quezon City, Philippines
- Novartis Investigative Site, Warsaw, Poland
- Romania (5):
  - Novartis Investigative Site, Cluj-Napoca, Jud Cluj
  - Novartis Investigative Site, Tg. Mures, Jud Mures
  - Novartis Investigative Site, Timișoara, Jud. Timis
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Iași
- Russia (3):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Voronezh
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A 1 arm study of valsartan but with 2 groups for analyses. The valsartan +antihypertensive group includes the patients who received background antihypertensive medication or received antihypertensive medication including amlodipine or HCTZ during the study.
Pre-assignment Details: These 2 groups were not randomized and considered to be 2 different populations since the patients in the valsartan+antihypertensive group had concomitant antihypertensive usage per individual patient's conditions at any time during treatment period.
Groups:
- CKD Patients: Valsartan + Antihypertensive Group: CKD Patients - Valsartan starting dose: ≥18 kg to <35 kg is 40 mg, ≥35 kg to <80 kg is 80 mg, ≥80 kg to ≤160 kg is 160 mg for 1 week then Valsartan maintenance dose: ≥18 kg to <35 kg is 80 mg, ≥35 kg to <80 kg is 160 mg, ≥80 kg to ≤160 kg is 320 mg after Week 8 if the Mean Sitting Systolic Blood Pressure (MSSBP) and/or Mean Sitting Diastolic Blood Pressure (MSDBP) was higher than 95th percentile for age, gender and height under the maintenance valsartan dose then add amlodipine and/or Hydrochlorothiazide (HCTZ). The valsartan +antihypertensive group includes patients who received background antihypertensive medication or received antihypertensive medication including amlodipine or HCTZ during the study.
- CKD Patients: Valsartan Alone: CKD Patients - Valsartan starting dose: ≥18 kg to <35 kg is 40 mg, ≥35 kg to <80 kg is 80 mg, ≥80 kg to ≤160 kg is 160 mg for 1 week then Valsartan maintenance dose: ≥18 kg to <35 kg is 80 mg, ≥35 kg to <80 kg is 160 mg, ≥80 kg to ≤160 kg is 320 mg.
- Non-CKD Patients: Valsartan + Antihypertensive Group: Non-CKD patients-Valsartan starting dose: ≥18 kg to <35 kg is 40 mg, ≥35 kg to <80 kg is 80 mg, ≥80 kg to ≤160 kg is 160 mg for 1 week then Valsartan maintenance dose: ≥18 kg to <35 kg is 80 mg, ≥35 kg to <80 kg is 160 mg, ≥80 kg to ≤160 kg is 320 mg after Week 8 if the Mean Sitting Systolic Blood Pressure (MSSBP) and/or Mean Sitting Diastolic Blood Pressure (MSDBP) was higher than 95th percentile for age, gender and height under the maintenance valsartan dose then add amlodipine and/or Hydrochlorothiazide (HCTZ). The valsartan +antihypertensive group includes patients who received background antihypertensive medication or received antihypertensive medication including amlodipine or HCTZ during the study.
- Non-CKD Patients: Valsartan Alone: Non-CKD patients-Valsartan starting dose: ≥18 kg to <35 kg is 40 mg, ≥35 kg to <80 kg is 80 mg, ≥80 kg to ≤160 kg is 160 mg for 1 week then Valsartan maintenance dose: ≥18 kg to <35 kg is 80 mg, ≥35 kg to <80 kg is 160 mg, ≥80 kg to ≤160 kg is 320 mg.
Period: Overall Study
Arm/Group | CKD Patients: Valsartan + Antihypertensive Group | CKD Patients: Valsartan Alone | Non-CKD Patients: Valsartan + Antihypertensive Group | Non-CKD Patients: Valsartan Alone
Started | 23 | 52 | 18 | 57
Completed | 16 | 37 | 14 | 50
Not Completed | 7 | 15 | 4 | 7
Not completed — Adverse Event | 6 | 9 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2 | 3
Not completed — Abnormal laboratory value(s) | 0 | 1 | 0 | 0
Not completed — Administrative problems | 0 | 1 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CKD Patients: Valsartan + Antihypertensive Group | CKD Patients: Valsartan Alone | Non-CKD Patients: Valsartan + Antihypertensive Group | Non-CKD Patients: Valsartan Alone | Total
Number analyzed (Participants) | 23 | 52 | 18 | 57 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.90 (3.35) | 12.30 (3.20) | 13.79 (2.64) | 14.37 (2.83) | 13.36 (3.130)
Age, Customized [Number; unit: participants]
  6 - 11 years | 10 | 22 | 3 | 10 | 45
  12 - 17 years | 13 | 30 | 15 | 47 | 105
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 3 | 20 | 51
  Male | 11 | 36 | 15 | 37 | 99

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) at End Point (Week 78 or Last Observation Carried Forward (LOCF)
Description: Sitting blood pressure was measured using a calibrated standard sphygmomanometer after the participants remained in sitting position for 5 minutes at clinic during the visit. The repeat sitting measurements were made at 2 to 3 minute intervals and the mean of three sSBP measurements were used as the average sitting office blood pressure for that visit.
Time Frame: Baseline, End Point (Week 78 or Last observation carried forward (LOCF)
Population: The Full Analysis set (FAS) included all patients who entered the treatment period. ) This OM looked at the Valsartan + Antihypertensive and Valsartan alone for ALL patients and did not break up the analysis between CKD and non-CKD patients.
Measure: Mean (Standard Deviation); unit: millimeter(s) of mercury (mmHg)
Groups:
- Valsartan + Antihypertensive Group: Valsartan starting dose: ≥18 kg to <35 kg is 40 mg, ≥35 kg to <80 kg is 80 mg, ≥80 kg to ≤160 kg is 160 mg for 1 week then Valsartan maintenance dose: ≥18 kg to <35 kg is 80 mg, ≥35 kg to <80 kg is 160 mg, ≥80 kg to ≤160 kg is 320 mg after Week 8 if the Mean Sitting Systolic Blood Pressure (MSSBP) and/or Mean Sitting Diastolic Blood Pressure (MSDBP) was higher than 95th percentile for age, gender and height under the maintenance valsartan dose then add amlodipine and/or Hydrochlorothiazide (HCTZ). The valsartan +antihypertensive group includes patients who received background antihypertensive medication or received antihypertensive medication including amlodipine or HCTZ during the study.
- Valsartan Alone: Valsartan starting dose: ≥18 kg to <35 kg is 40 mg, ≥35 kg to <80 kg is 80 mg, ≥80 kg to ≤160 kg is 160 mg for 1 week then Valsartan maintenance dose: ≥18 kg to <35 kg is 80 mg, ≥35 kg to <80 kg is 160 mg, ≥80 kg to ≤160 kg is 320 mg.
Arm/Group | Valsartan + Antihypertensive Group | Valsartan Alone
Number analyzed (Participants) | 41 | 109
millimeter(s) of mercury (mmHg) | -13.3 (13.69) | -15.5 (13.35)

2. Secondary Outcome: Number of Participants With MSSBP, MSDBP and (MSSBP and MSDBP Combined) < 95th Percentile for Gender, Age, and Height
Description: Number of Participants with Mean sitting systolic (MSSBP) and mean sitting diastolic(MSDBP) blood pressure and both combined less than the 95th percentile for age, gender and height
Time Frame: End Point (Week 78 or Last observation carried forward (LOCF)
Population: The Full Analysis set (FAS) included all patients who entered the treatment period. This analysis includes only participants with baseline MSSBP or MSDBP or (MSSBP or MSDBP combined) ≥95th percentile for gender, age and height. n analyzed is displayed in left column. This OM did not break up the analysis between CKD and non-CKD patients.
Measure: Number; unit: Number of Participants
Arm/Group | Valsartan + Antihypertensive Group | Valsartan Alone
Number analyzed (Participants) | 41 | 109
Number of Participants
  MSSBP (n=39, 105) | 23 | 90
  MSDBP (n=28, 51) | 20 | 47
  MSSBP and MSDBP combined (n=40, 105) | 22 | 88

3. Secondary Outcome: Percentage of Chronic Kidney Disease (CKD) Patients Who Had >=50% Reduction in Urine Albumin/Creatinine Ratio (UACR) From Baseline to End Point
Description: Percentage of Patients with CKD who had Urine albumin creatinine reduction >/= 50% from baseline
Time Frame: Baseline, End Point (Week 78 or Last observation carried forward (LOCF)
Population: The Safety set (SAF) included all patients who received at least one dose of study medication that has Chronic Kidney Disease (CKD) only
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan + Antihypertensive Group | Valsartan Alone
Number analyzed (Participants) | 23 | 52
Percentage of patients | 50.0 (404.08) | 41.9 (138.66)

4. Primary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (MsDBP) at End Point (Week 78 or Last Observation Carried Forward (LOCF)
Description: Sitting blood pressure was measured using a calibrated standard sphygmomanometer after the participants remained in sitting position for 5 minutes at clinic during the visit. The repeat sitting measurements were made at 2 to 3 minute intervals and the mean of three sDBP measurements were used as the average sitting office blood pressure for that visit.
Time Frame: Baseline, End Point (Week 78 or Last observation carried forward (LOCF)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeter(s) of mercury (mmHg)
Arm/Group | Valsartan + Antihypertensive Group | Valsartan Alone
Number analyzed (Participants) | 41 | 109
millimeter(s) of mercury (mmHg) | -10.3 (11.94) | -10.8 (11.45)

5. Secondary Outcome: Percentage of Chronic Kidney Disease (CKD) Patients Who Had Estimated Glomerular Filtration Rate (eGFR) Decrease > 25 % From Baselinefrom Baseline to End Point
Description: Percentage of Patients with CKD who had eGFR decrease > 25 % from Baseline
Time Frame: Baseline, End Point (Week 78 or Last observation carried forward (LOCF)
Population: The Safety set (SAF) included all patients who received at least one dose of study medication.that has Chronic Kidney Disease (CKD)
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan + Antihypertensive Group | Valsartan Alone
Number analyzed (Participants) | 23 | 52
Percentage of patients | 30.4 (404.08) | 27.5 (138.66)

ADVERSE EVENTS:
Arm/Group | Valsartan + Antihypertensive Group | Valsartan Alone | CKD Patients: Valsartan + Antihypertensive Group | CKD Patients: Valsartan Alone | Non-CKD Patients: Valsartan + Antihypertensive Group | Non-CKD Patients: Valsartan Alone
Serious Adverse Events (participants affected / at risk) | 8/41 | 7/109 | 7/23 | 4/52 | 1/18 | 3/57
Other Adverse Events (participants affected / at risk) | 34/41 | 68/109 | 18/23 | 36/52 | 16/18 | 32/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan + Antihypertensive Group (N=41) | Valsartan Alone (N=109) | CKD Patients: Valsartan + Antihypertensive Group (N=23) | CKD Patients: Valsartan Alone (N=52) | Non-CKD Patients: Valsartan + Antihypertensive Group (N=18) | Non-CKD Patients: Valsartan Alone (N=57)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Oesophageal polyp (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Drug abuse (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0
IgA nephropathy (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Lupus nephritis (Renal and urinary disorders) | 3 | 1 | 3 | 1 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan + Antihypertensive Group (N=41) | Valsartan Alone (N=109) | CKD Patients: Valsartan + Antihypertensive Group (N=23) | CKD Patients: Valsartan Alone (N=52) | Non-CKD Patients: Valsartan + Antihypertensive Group (N=18) | Non-CKD Patients: Valsartan Alone (N=57)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Myopia (Eye disorders) | 1 | 1 | 0 | 0 | 1 | 1
Retinal vascular disorder (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 2 | 0 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 7 | 2 | 4 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 5 | 2 | 2 | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 8 | 1 | 5 | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 3 | 2 | 2 | 0 | 1
Toothache (Gastrointestinal disorders) | 3 | 1 | 2 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 5 | 4 | 4 | 3 | 1 | 1
Asthenia (General disorders) | 2 | 1 | 1 | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 12 | 18 | 8 | 12 | 4 | 6
Acarodermatitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0
Enterobiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 3 | 1 | 1 | 0 | 2 | 1
Mycoplasma infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 11 | 22 | 7 | 14 | 4 | 8
Pharyngitis (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 4 | 1 | 0 | 1 | 4
Rhinitis (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 17 | 1 | 12 | 1 | 5
Urinary tract infection (Infections and infestations) | 2 | 3 | 2 | 2 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 4 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 3 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 8 | 17 | 4 | 6 | 4 | 11
Headache (Nervous system disorders) | 14 | 23 | 8 | 11 | 6 | 12
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 18 | 12 | 12 | 6 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 1 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 1 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3 | 2 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 1 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 3 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 2 | 2 | 2 | 0 | 0
Pallor (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single- site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.